CLINICAL TRIAL: NCT04881149
Title: Rollover Study to Evaluate Histological Results of Radiofrequency Device Treatments on the Flanks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN20-FIRM-LIPO-ROLLOVER
Record Dates: First submitted 2021-05-04; First posted 2021-05-11 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All Study Participants (Experimental): The TempSure will be used on the flanks during this study. Subjects will receive 1 biopsy in the treatment area on the flank. Subjects will also receive 1 biopsy sample on the contralateral side, where they did not receive treatment. Each subject had 1 control sample (tissue that was taken from an area where no treatment was received), and 1 treatment sample (tissue taken from an area that had been subjected to the treatment).
  Interventions: Device: TempSure treatment

INTERVENTIONS:
Device: TempSure treatment — Self-controlled, single-arm study using the TempSure device.

SUMMARY:
The purpose of this study is to evaluate histological results of the treatments with the TempSure Firm handpiece on the flanks performed in the CYN20-FIRM-LIPO study.

DETAILED DESCRIPTION:
Up to 10 subjects will be enrolled at up to 3 study centers. Subjects will receive 2 biopsies, 1 biopsy in the treatment area (the flanks) and 1 biopsy outside of the treatment area to serve as a control.

ELIGIBILITY:
Inclusion Criteria:

• Subject has completed their participation in the CYN20-FIRM-LIPO study.

Exclusion Criteria:

* The subject has not had any other treatment in the treatment area after their involvement in the CYN20-FIRM-LIPO study.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (1):
- JUVA Skin & Laser Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: biopsy samples
Period: Overall Study
Arm/Group | All Study Participants
Started | 7; 14 biopsy samples
Control Biopsy | 7; 7 biopsy samples
Treatment Biopsy | 7; 7 biopsy samples
Completed | 7; 14 biopsy samples
Not Completed | 0; 0 biopsy samples

BASELINE CHARACTERISTICS:
Population: This study is described as only being composed of 1 arm because every subject underwent the same treatment procedure and had a control biopsy taken (in an area that was not treated) to be compared to the treatment biopsy.
Groups:
- TempSure Device: The TempSure will be used on the flanks during this study.
  TempSure treatment: Self-controlled, single-arm study using the TempSure device.
Arm/Group | TempSure Device
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 2
  African American | 1
  Caucasian | 4
FitzPatrick Skin Type [Count of Participants; unit: Participants] — Measure Description: The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes used is cited in the reference section.
  Participants
    FitzPatrick Skin Type I | 0
    FitzPatrick Skin Type II | 0
    FitzPatrick Skin Type III | 1
    FitzPatrick Skin Type IV | 4
    FitzPatrick Skin Type V | 1
    FitzPatrick Skin Type VI | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Samples With Different Levels of Elastin When Compared to Baseline Samples From the Same Patient
Description: Sections of skin were removed using the punch biopsy technique to render a microscopic diagnosis. Each specimen was preserved with a fixative and then stained using Hemotoxylin & Eosin, Verhoeff and Masson Red/Fast Green and/or nitroblue tetrazolium chloride (NBTC) staining methods. If using Hemotoxylin & Eosin, Verhoeff and Masson Red/Fast Green staining, samples were assessed and evaluated by the amount of elastin. If using NBTC staining, samples were assessed and evaluated to differentiate between the blue-stained viable cells and the unstained thermally damaged cells. The samples were examined by a qualified pathologist. The visual changes between the treated samples and the control samples were examined, with no typical unit of measure used to quantify the difference. Simply, control and treatment images were compared to each other with a qualitative analysis of the changes. The number of samples with different levels of elastin (control compared to treatment) is reported.
Time Frame: 1 Week (7-10 days) Post Baseline
Measure: Number; unit: biopsy samples
Units Other Than Participants: biopsy samples
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Number analyzed (biopsy samples) | 14
biopsy samples | 0

2. Primary Outcome: Number of Treatment Samples With Different Levels of Dermis Collagen When Compared to Baseline Samples Taken From the Same Patient
Description: Sections of skin were removed using the punch biopsy technique to render a microscopic diagnosis. Each specimen was preserved with a fixative and then stained using Hemotoxylin & Eosin, Verhoeff and Masson Red/Fast Green and/or nitroblue tetrazolium chloride (NBTC) staining methods. If using Hemotoxylin & Eosin, Verhoeff and Masson Red/Fast Green staining, samples were assessed and evaluated by the amount of collagen. If using NBTC staining, samples were assessed and evaluated to differentiate between the blue-stained viable cells and the unstained thermally damaged cells. The samples were examined by a qualified pathologist. The visual changes between the treated samples and the control samples were examined, with no typical unit of measure used to quantify the difference. Simply, control and treatment images were compared to each other with a qualitative analysis of the changes. The number of samples with different levels of collagen (control compared to treatment) is reported.
Time Frame: 1 Week (7-10 days) Post Baseline
Measure: Number; unit: biopsy samples
Units Other Than Participants: biopsy samples
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Number analyzed (biopsy samples) | 14
biopsy samples | 0

ADVERSE EVENTS:
Time Frame: All adverse events were followed through study completion, an average of 7 months.
Groups:
- Treatment Flank: The TempSure was used on the flanks during this study. Subjects receive 1 biopsy in the treatment area on the flank. Each subject had 1 treatment sample (tissue taken from an area that had been subjected to the treatment).
- Control Flank: Subjects receive 1 biopsy sample on the contralateral side, where they did not receive treatment.
Arm/Group | Treatment Flank | Control Flank
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Flank (N=7) | Control Flank (N=7)
Pain/tenderness (Nervous system disorders) | 1 | 0
Irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Scabbing (Skin and subcutaneous tissue disorders) | 1 | 1
Bruising (Skin and subcutaneous tissue disorders) | 2 | 1
Itching (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT04881149/Prot_001.pdf